CLINICAL TRIAL: NCT02651337
Title: Quantitative Characterization of Safe Irrigation for Ventricular Shunt Catheters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcyone Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P000009795
Record Dates: First submitted 2015-12-21; First posted 2016-01-11 (Estimated); Results first posted 2020-09-21 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-08

CONDITIONS: Hydrocephaly
MeSH Terms: conditions — Hydrocephalus | interventions — Drainage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Drainage with Alivio in-line Flusher (Experimental): Volume of saline needed to drain CSF using the Alivio in-line Flusher historically compared with volume of saline needed to drain CSF using a standard syringe
  Interventions: Device: Cerebrospinal Fluid (CSF) Drainage

INTERVENTIONS:
Device: Cerebrospinal Fluid (CSF) Drainage — Placement of Alivio in line flusher during CSF drainage
  Other Names: Alivio in line flusher

SUMMARY:
The objective of this pilot study is to perform a set of pressure and flow rate measurements in order to quantitatively characterize safe irrigation or "flushing" of a ventricular shunt catheter, a routine maneuver performed by a neurosurgeon during a shunt revision surgery. This maneuver involves injecting saline with a syringe to clear plugged shunt catheters. Based on data obtained in Stage I of the study, a device has been fabricated which provides the same small-volume pulse of fluid used by surgeons. In Stage II of the study, pressure and flow rate measurements generated by this specialized flusher device will be collected and measured.

DETAILED DESCRIPTION:
Primary Objective: To collect pressure and flow rate measurements during shunt revision surgeries in human patients.

Pressure recordings of the injected fluid will be obtained using disposable off-the-shelf sterile pressure transducers (which are typically used for intracranial and arterial pressures monitoring) readily available in the operating room. First, the surgeon will attempt to flush the catheter using the Alcyone in-line Flusher device. If this fails, the surgeon may elect to attempt to flush using a standard syringe attached to the catheter. The flow rates will be measured by video, recording the syringe during the flushing maneuver, and then extracting plunger motion information by applying image processing on the acquired videos. In the event the recording equipment is not available (in that these operations are usually unscheduled and sometimes urgent), the same irrigation techniques may be used without the pressure recordings.

Secondary Objective: To analyze the collected data and establish maximal allowable injection pressure and flow rate. The collected data segments for each patient will be analyzed and maximal values for pressure and the saline injection rate will be recorded in a spreadsheet. Inter-patient variation in the results, presumably due to different degrees of occlusion, will be statistically evaluated. We will also determine if any of the catheters which appear occluded in the operating room resume flow with the flushing maneuvers.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be 30 days to 35 years of age, of any race or gender.
2. Subjects must be scheduled to undergo a neurosurgical procedure potentially requiring a revision of neurosurgical catheters.
3. Subjects aged >18 years of age must be willing and able to provide written informed consent. Parental consent will be required for minors.

Exclusion Criteria:

1. Inability or unwillingness of subject or parent/guardian to give informed consent/assent.
2. Judgment of the investigator, surgeon, or any member of the care team (including anesthesiology or operating room nursing staff) that participation in the study will interfere with, or be detrimental to, administration of optimal healthcare of the subject.
3. Inability or unwillingness of subject to endure the test or any other condition that would preclude or bias the results of the study according to the judgment of the investigator.

Ages: 30 Days to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2016-06-04 (Actual); Study Completion 2016-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Warf, MD Warf, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Boop FA, Medhkour A, Honeycutt J, James C, Cherny WB, Duntsch C. In vitro testing of current spread during ventricular catheter coagulation using diathermy. Technical note. J Neurosurg. 2007 Feb;106(2 Suppl):165-8. doi: 10.3171/ped.2007.106.2.165. PMID 17330548
- [Result] Naradzay JF, Browne BJ, Rolnick MA, Doherty RJ. Cerebral ventricular shunts. J Emerg Med. 1999 Mar-Apr;17(2):311-22. doi: 10.1016/s0736-4679(98)00168-1. PMID 10195493
- See also: Book Chapter: ISBN13: 9781588905109 — http://link.springer.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 5 participants consented for study participation, 4 patients were enrolled
Period: Overall Study
Arm/Group | Drainage With Alivio In-line Flusher
Started | 5
Completed | 4
Not Completed | 1

BASELINE CHARACTERISTICS:
Population: Consent was received by five (5) subjects, whom completed baseline assessments; only four (4) subjects participated in the study.
Arm/Group | Drainage With Alivio In-line Flusher
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3
  Between 18 and 65 years | 2
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 15 [1 to 27]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: To Demonstrate That the Flusher Can be Primed, Connected, and Activated in a Sterile Clinical Setting Per the Instructions for Use by the Treating Investigator .
Description: Criteria for success:
  Investigator Determination if the Flusher can be properly primed. Investigator Determination if the Flusher can be easily connected to current shunt components.
  Investigator Determination if the Flusher can be activated.
  The following scenarios were also assessed:
  A noticeable resistance to compression/collapse of the dome to indicate that the Ventricular Catheter is too tightly blocked to be flushed.
  If the dome does not refill the Ventricular Catheter may still be non-flowing. If the dome refills, the flushing procedure may be repeated as needed and/or as determined reasonable by the surgeon.
Time Frame: Intra-procedural
Measure: Count of Participants; unit: Participants
Groups:
- Alivio Ventricular Flusher Device: The Alivio Ventricular Flusher Device (Flusher) is used in the treatment of patients with hydrocephalus. It is an accessory component that may be connected to a shunt system, which is designed to aid in resuming flow in a non-flowing ventricular catheter.
Arm/Group | Alivio Ventricular Flusher Device
Number analyzed (Participants) | 4
Participants
  Ability to Prime the Flusher | 4
  Adequate Flusher Connection to Shunt | 4
  System Flushed by dome compression | 4
  Dome able to be Refilled | 4
  Dome able to be Evacuated | 3
Statistical Analysis 1: Comparison: Alivio Ventricular Flusher Device; Test type: Other — It is a one arm clinical study. No comparison between groups was made; The study tested the hypothesis that the Alivio flusher could increase flow in occluded or sluggish flowing catheters. Analysis was made on the basis of the procedural results related to priming the flusher, connecting the flusher to the shunt, flushing the system by dome compression, the ability to refill the dome, and the ability to evacuate the dome

ADVERSE EVENTS:
Arm/Group | Drainage With Alivio In-line Flusher
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No